CLINICAL TRIAL: NCT06873633
Title: A Phase II Study to Evaluate the Safety, Pharmacokinetics, Antiviral Activity and Acceptability of Remdesivir (VEKLURY®) in Hospitalized Children Aged 0 to Less Than 2 Years With Respiratory Syncytial Virus (RSV)-Associated Lower Respiratory Tract Infection.
Brief Title: Safety, Pharmacokinetics, and Antiviral Activity of Remdesivir (VEKLURY®) in Hospitalized Children With RSV
Acronym: THAI-CARES RSV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: AMS-PHPT Research Collaboration (Unknown); Chiang Mai University (Other); Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THAI-CARES RSV; CO-US-540-7443 (Other Grant/Funding Number: Gilead)
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: respiration disorders; RSV infection; Respiratory Syncytial Virus Hospitalizations
MeSH Terms: conditions — Respiration Disorders; Respiratory Syncytial Virus Infections | interventions — remdesivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (control arm). (No Intervention): Standard of care treatments will be delivered according to local practice at each hospital. The standard of care for lower respiratory tract infection includes oxygen therapy as needed, bronchodilators, intravenous fluids, in some cases the use of steroids, antibiotics and any treatment for underlying disease.
- Intervention arm (Experimental): Remdesivir will be used in combination with the standard of care. Remdesivir will be administered by intravenous infusion every 24 hours for five (5) consecutive days with a dosage based on the participant's weight at the time of the randomisation.
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Remdesivir — Remdesivir (RDV) has shown potent antiviral activity against RSV A in an animal model. Remdesivir has been also shown to be a safe treatment option in pediatric patients hospitalized with COVID-19. Based on previous clinical evidence and preclinical data, to address the unmet medical need for safe and effective RSV therapy, this study is being conducted to investigate remdesivir in infants and children (aged 0 days to <2 years) as a potential treatment for RSV infection.
  Other Names: VEKLURY®
  Arms: Intervention arm

SUMMARY:
THAI-CARES RSV Study is a Phase II, open-label, multicenter, randomized controlled trial with a two-arm, parallel-group design. The study aims to assess the safety, efficacy, and acceptability of a five-day course of Remdesivir (VEKLURY®) in children under two years of age who are hospitalized with confirmed respiratory syncytial virus (RSV) infection, as determined by either a rapid antigen test or RT-PCR. The primary objectives include evaluating the treatment's safety profile, its ability to significantly reduce RSV replication, and its overall acceptance in this patient population.

DETAILED DESCRIPTION:
An overall target of 120 participants will be involved in the study. Eligible participants will be randomized (1:1) to receive ARM 1: Standard of care alone (control arm). ARM 2: Remdesivir in combination with the standard of care. Remdesivir will be administered by intravenous infusion every 24 hours for five (5) consecutive days. Each participant will be followed during hospitalization plus 7-10 days after Day 6* for final visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parents/caregivers
* Aged 0 to <2 years
* Weighing at least 2.0 kg
* Onset of RSV associated-symptoms within 1 week of screening
* Confirmed* with RSV infection (by rapid antigen test or RT PCR)
* Hospitalized children fulfilling at least two of the following three RSV disease severity criteria:

  * Inadequate oral feeding
  * Inadequate oxygen saturation (peripheral capillary oxygen saturation [SpO2] <95% on room air or requiring oxygen supplementation to maintain SpO2 ≥95%)
  * Signs of respiratory distress (respiratory rate of ≥60 breaths per min for children aged up to 1 year, or ≥40 breaths per min for those older than 1 year, or accessory respiratory muscles use [subcostal, intercostal, or suprasternal retraction], or both)

Exclusion Criteria:

* Preterm infants (gestational age at birth less than 37 weeks) who are aged <56 days
* Being hospitalized for other clinically relevant concurrent conditions (except for risk factors for severe RSV, e.g., cardiac disease, pulmonary disease, genetic disease, and prematurity)
* Concurrent treatments with other agents with actual or possible direct antiviral activity against RSV <24 hours prior to study drug dosing (e.g. ribavirin)
* ALT or AST > 5 × ULN
* eGFR <30 mL/min/1.73m2 using the Schwartz formula if aged ≥1 year; or if aged <1 year based on a creatinine value cut off dependent on chronological age
* Any major congenital renal anomaly if <28 days
* Apgar score < 5 when last recorded if age <24 hours
* Known hypersensitivity to the study drug, the metabolites, or formulation excipient.
* On renal replacement therapies (e.g., intermittent hemodialysis, peritoneal dialysis, continuous renal replacement therapy)
* Any condition that, in the opinion of the site investigator, would make participation in the study unsafe for the child, or comprise the study objectives

Ages: 0 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of Remdesivir | 1 Week
  Outcome Measures:
  Occurrence of the following events from the time of randomization until the last study visit:
  * serious adverse events (SAEs);
  * adverse events (AEs) of Grade 3 or higher
  * treatment-related AEs
  * AEs leading to treatment discontinuation
  * treatment-related AEs leading to treatment discontinuation
  * AEs of Grade 3 or higher leading to treatment discontinuation
  Acceptability of daily remdesivir infusions to children, health care personnel, and caregivers assessed through questionnaires and direct observation.

SECONDARY OUTCOMES:
Evaluation of the RSV RNA viral load | 1 Week
  Outcome measures:
  * Reduction in RSV RNA viral load reduction from Day 1 to Day 6, i.e. one day after the end of treatment.
  * Time from Day 1 to RSV RNA viral load drop below the RT-PCR quantification limit until Day 6.
  * Area under the RSV RNA viral load-time curve (AUC) from Day 1 until Day 6.
Efficacy of Remdesivir | 1 Week
  Ourtome Measures:
  Improvement on the PRESS 6-step ordinal scale from Day 1 until Day 6. PK parameters will be estimated for remdesivir and its metabolites GS-704277 and GS-44152417.

CONTACTS AND LOCATIONS:
Overall Officials: Tim R Cressey, Principal Investigator — AMS-PHPT Research Collaboration, Faculty of Associated Medical Sciences, Chiang Mai University; Tavitiya Sudjaritruk, Principal Investigator — Department of Pediatrics, Faculty of Medicine, Chiang Mai University; Pablo Rojo, Principal Investigator — Hospital Materno Infantil 12 de Octubre
Locations (8):
- Thailand (8):
  - Center of Excellence for Pediatric Infectious Diseases and Vaccines Faculty of Medicine, Chulalongkorn University (CE-PID), Bangkok
  - Nakornping Hospital, Chiang Mai
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Khon Kaen Hospital, Khon Kaen
  - Lampang Hospital, Lampang
  - Mahasarakham Hospital, Maha Sarakham
  - Samut Sakhon Hospital, Samut Sakhon

IPD SHARING:
Plan to Share IPD: No